CLINICAL TRIAL: NCT00796341
Title: Does Endometrial Injury in the Non-Transfer Cycle Improve the IVF-ET Outcome in the Subsequent Cycle in Patients With Previous Failed IVF Cycles: A Randomized Control Trial
Brief Title: Endometrial Injury and IVF-ET Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangalore Assisted Conception Centre (Other)
Responsible Party: Dr Kamini A Rao, Bangalore Assisted Conception Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: endometrial injury study
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-11

CONDITIONS: Infertility
Keywords: invitro-fertilization ,embryo transfer,endometrial injury
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: PIPELLE ENDOMETRIAL SAMPLING
- 2 (No Intervention)

INTERVENTIONS:
Procedure: PIPELLE ENDOMETRIAL SAMPLING — Pipelle endometrial sampling will be done twice between 7th to 10th day and 24th to 26th d in the cycle prior to IVF.
  Other Names: Endometrial sampling
  Arms: 1

SUMMARY:
Implantation of the human embryo is the limiting factor in the success of invitro-fertilization and embryo transfer(IVF-ET).We wanted to find out whether creating a local injury to the endometrium in the non-transfer cycle would improve the IVF-ET outcome in the subsequent cycle.We believe that the injury created causes release of substances which help in implantation.

DETAILED DESCRIPTION:
Study Design and Subjects: This is a randomized control study designed to evaluate the effect of local injury to the endometrium in non-transfer cycle in patients with previous failed IVF.

Patients will be randomly allotted to control and intervention group The patients in the intervention group Pipelle endometrial sampling 7-10th day and 24-26th day in the cycle prior to IVF transfer cycle.

Outcome Measures: Clinical pregnancy rate,implantation rate and ongoing pregnancy rate.

SAMPLE SIZE: 100 PATIENTS (50 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Previous failed In-vitro fertilization embryo transfer cycle
* Patients who are good responders and have good quality embryos in the previous attempts
* Age of patients upto 37yrs

Exclusion Criteria:

* Those detected to have endometrial tuberculosis in the past, including those treated with Antituberculosis treatment
* Those with intramural fibroid distorting the endometrial cavity/sub-mucous myoma
* Those with sonographically detected hydrosalpinx

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
PRIMARY OUTCOME MEASURE:IMPLANTATION RATE; | 9 MONTHS

SECONDARY OUTCOMES:
CLINICAL PREGNANCY RATE,ONGOING PREGNANCY RATE | 9 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: SACHIN A NARVEKAR, MD, Principal Investigator — Bangalore Assisted Conception Centre
Locations (1):
- Bangalore Assisted Conception Centre, Bangalore, Karnataka, India

REFERENCES:
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877
- [Derived] Lensen SF, Armstrong S, Gibreel A, Nastri CO, Raine-Fenning N, Martins WP. Endometrial injury in women undergoing in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Jun 10;6(6):CD009517. doi: 10.1002/14651858.CD009517.pub4. PMID 34110001